CLINICAL TRIAL: NCT01818349
Title: Gait Performance and Lower-limb Muscle Strength Improved in Both Upper-limb and Lower-limb Isokinetic Training Programs in Individuals With Chronic Stroke
Brief Title: Impact of Training on Gait and Strength in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-hélène Milot, professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRSC-44059
Record Dates: First submitted 2013-03-15; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Stroke
Keywords: stroke; exercise; muscle strength; gait; rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- isokinetic lower-limb training (Active Comparator): 3 times/week for 6 weeks
  Interventions: Other: isokinetic lower-limb training
- isokinetic uppe-limb training (Placebo Comparator): 3 times/week for 6 weeks
  Interventions: Other: isokinetic upper-limb training

INTERVENTIONS:
Other: isokinetic lower-limb training — concentric training of the affected plantarflexors, hip flexors and hip extensors
  Arms: isokinetic lower-limb training
Other: isokinetic upper-limb training — concentric training of the affected wrist extensors, elbow flexors and shoulder flexors
  Arms: isokinetic uppe-limb training

SUMMARY:
Background: A discrepancy between strength gain and gait changes following various training programs aimed at improving gait function after stroke has been noted. A mismatch between the training program and gait parameters could explain this finding.

Objective: To evaluate the impact of an isokinetic-strengthening program, matching the requirements of the affected lower-limb muscle groups involved in the energy generation of gait, to a control intervention, on gait performance and muscle strength.

Hypothesis: The isokinetic training program of the affected lower-limb muscles would produce greater changes in gait performance and strength than a control intervention not aiming at training these muscle groups.

Design: Single-blinded randomized controlled trial.

Participants: A convenient sample of 30 individuals with chronic hemiparesis.

Interventions: Participants were randomly assigned into two groups (n=15), each training three times/week for six weeks. The experimental group trained the affected plantarflexors, hip flexors and extensors concentrically, while the control group trained the affected upper-limb muscles.

Main outcome measures: Baseline values and post-training values, taken at the end of the training program, of maximal voluntary concentric strength, gait speed and peak positive power.

ELIGIBILITY:
Inclusion Criteria:

* have a chronic (six months or more) unilateral stroke
* be able to walk 10 meters independently with or without a cane
* present residual weakness at the affected lower limb
* have an activity tolerance of at least two hours with a rest period

Exclusion Criteria:

* receptive aphasia
* incontinence
* unstable medical condition
* history of injury
* anesthesia at the lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-03; Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
change in gait speed | gait speed was assessed at baseline and at the completion of the 6-week training (i.e. week #7)
  change in gait speed, in meter/second, was assessed as the difference between the baseline and week #7 values.
change in peak positive power | peak positive power was assessed at baseline and at the completion of the 6-week training (i.e. week #7)
  peak positive power was evaluated at the affected plantarflexors, hip flexors and hip extensors. Also, change in peak positive power, in weight/kilogram, was assessed as the difference between the baseline and week #7 values.

SECONDARY OUTCOMES:
change in maximal voluntary concentric strength | maximal voluntary concentric strength was assessed at baseline and at the completion of the 6-week training (i.e. week #7)
  maximal voluntary concentric strength was evaluated at the affected plantarflexors, hip flexors and hip extensors. Also, change in maximal voluntary concentric strength, in Newton-metre, was assessed as the difference between the baseline and week #7 values.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Nadeau, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Institut de réadaptation Gingras-Lindsay, Montreal, Quebec, Canada